CLINICAL TRIAL: NCT05089721
Title: Questionnaire for Evaluation of Uterotonic Usage Habits of Obstetricians and Anesthesiologist
Brief Title: Questionnaire for Obstetricians and Anesthesiologist
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Selin Erel, Assistant Professor in Department of Anesthesiology and Reanimation, Gazi University
Other Study IDs: ecd9b925a955474783d32b99b7f21
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-01

CONDITIONS: Uterine Bleeding; Atony, Uterine; Cesarean Section Complications
MeSH Terms: conditions — Uterine Hemorrhage; Uterine Inertia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Anesthesiologist
- Obstetricians

SUMMARY:
The research was planned as a face-to-face survey evaluation. The questionnaire will be applied to obstetricians and anesthesiologists working in public and private hospitals. The universe of the research will be selected by simple random sampling method, and the total number of people who will participate is planned to be 200, approximately 100 from each of the two branches. Our survey consists of 5 parts structurally. Demographic data, rate of cesarean section and postpartum hemorrhage, uterotonic agent preferences in low/high risk cesarean section surgeries, the preference for second-line uterotonic agents, and the dose preferences of uterotonic agents.

ELIGIBILITY:
Inclusion Criteria: obstetricians and anesthesiologists who want to participate in the survey

Exclusion Criteria: the ones who do not want to participate

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Through national obstetrics and anesthesiologist associations, the survey will be sent to the participant's e-mail addresses. Those who answer the questionnaire will be included in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-21 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Uterotonic usage habits in postpartum hemorrhage | 3 months
  to learn the uterotonic use preferences of both obstetricians and anesthesiologists in postpartum

SECONDARY OUTCOMES:
Uterotonic usage habits in elective cesearean section | 3 months
  to learn the uterotonic use preferences of both obstetricians and anesthesiologists in elective cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University School of Medicine, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
overall results of survey will be shared, individual answers of participants wont be shared